CLINICAL TRIAL: NCT00678093
Title: The Effects of the Mulligan Mobilisation Sustained Natural Apophyseal Glide (SNAG) in the Lumbar Flexion Range of Asymptomatic Subjects as Measured by the Zebris CMS20 3-D Motion Analysis System
Brief Title: Effects of a Mulligan Mobilisation in the Lumbar Flexion Range of Asymptomatic Subjects
Acronym: Mulligan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Evdokia Billis, Lecturer in Physiotherapy, Department of Physiotherapy, TEI of Lamia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mulligan
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Low Back Pain
Keywords: Low back pain; Manual therapy; Mulligan snag
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNAG (Experimental): SNAG is a painless and gentle manual technique, mimicking a slide with concurrent active movement, performed in the lumbar spine (in this study) by an experienced manual therapist-physiotherapist.
  Interventions: Other: Application of the SNAG technique

INTERVENTIONS:
Other: Application of the SNAG technique — SNAG is a painless and gentle manual technique, mimicking a slide with concurrent active movement, performed in the lumbar spine (in this study) by an experienced manual therapist-physiotherapist.
  Other Names: Sustained Natural Apophyseal Glide; Mulligan mobilisation

SUMMARY:
Mulligan's mobilisation techniques are believed to increase the range of movement (ROM) in patients with low back pain. The primary aim of this study was to investigate the mechanical effects of Mulligan's "SNAG" technique on lumbar flexion ROM. The secondary aim was to measure the intra- and inter-day reliability of lumbar ROM employing the same procedure, and utilising a 3-D motion analysis system for measuring range of motion (ROM).

DETAILED DESCRIPTION:
The primary aim of this study was to investigate the mechanical effects of Mulligan's "SNAG" technique on lumbar flexion ROM. The secondary aim was to measure the intra- and inter-day reliability of lumbar ROM employing the same procedure. For the interventional component of the study, 49 asymptomatic volunteers participated in it. Subjects were randomly assigned into either a treatment (SNAG) group (n=25), or a placebo (SHAM) group (n=24). The "SNAG" technique was applied on L3 and L4 spinal levels by an experienced manual therapist. SNAGs were performed with active flexion in sitting, 10 times at each level. The placebo-SHAM was similar to the SNAG without however applying the appropriate direction or force. Lumbar ROM was measured by a three dimensional electronic goniometer (Zebris CM20), before and after each technique. For the reliability component, five measurements in two different days (one week apart) were performed in 20 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic
* health individuals

Exclusion Criteria:

* Low back pain
* spinal pathology
* vascular or heart problems
* subjects taking anticoagulants

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Range of Movement (ROM) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Billis, MSc, Principal Investigator — University of Manchester
Locations (1):
- Centre for Rehabilitation Science, Manchester, United Kingdom

REFERENCES:
- [Derived] Moutzouri M, Billis E, Strimpakos N, Kottika P, Oldham JA. The effects of the Mulligan Sustained Natural Apophyseal Glide (SNAG) mobilisation in the lumbar flexion range of asymptomatic subjects as measured by the Zebris CMS20 3-D motion analysis system. BMC Musculoskelet Disord. 2008 Oct 1;9:131. doi: 10.1186/1471-2474-9-131. PMID 18828921